CLINICAL TRIAL: NCT04319081
Title: Multicenter, Observational and Prospective Study to Evaluate Changes in Cognitive Function in Patients Treated With PCSK9 Inhibitors (MEMOGAL)
Brief Title: Study to Evaluate Changes in Cognitive Function in Patients Treated With PCSK9 Inhibitors
Acronym: MEMOGAL
Status: Completed | Type: Observational
Sponsor: Jose Seijas Amigo (Other)
Responsible Party: Sponsor-Investigator, Jose Seijas Amigo, Pharmacist, Hospital Clinico Universitario de Santiago
Organization: Hospital Clinico Universitario de Santiago (Other)
Other Study IDs: JSA-ALI-2019-01; 2019/653 (Other: CEIm-G); PMID: 33941059 (Other: pubmed)
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Function; Hypercholesterolemia; Quality of Life
Keywords: Cognitive Function; Hypercholesterolemia; Quality of Life; Pharmacoeconomics; PCSK9 inhibitors; Alirocumab; Evolocumab
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uncontrolled patients with hypercholesterolemia: Patients that meet criteria inclusions and they have just started to take Alirocumab or Evolocumab
  Interventions: Drug: PCSK9 inhibitor

INTERVENTIONS:
Drug: PCSK9 inhibitor — Patients are included after PCSK9 inhibitors prescription , at the first dispensation

SUMMARY:
The main objective will be to evaluate the changes in the cognitive function in naive patients treated with PCSK9 inhibitors (Alirocumab and Evolocumab) by using the Montreal Cognitive Assesment questionnaire (MOCA).

The secondary objectives will be: 1) To evaluate the levels of LDL-cholesterol changes from the beginning to the end of the study 2) To evaluate changes in Quality of Life among the EuroQol EQ-5D-3L questionnaire (it will also be associated to the cognitive function) 3) Assesment of direct costs in medications and outpatients consultations related with the health procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or over
* To start with the first funded dose of PCSK9 inhibitors ( LDL > 100 mg/dL)
* Maximum dose or statin intolerance

Exclusion Criteria:

* Diagnosis of any disease related with cognitive deterioration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with familial hypercholesterolemia (homozygous and heterozygous) and/or cardiovascular disease with LDL-cholestrol value > 100 mg/dL and maximum statine doses or intolerance. With a first prescription of PCSK9 inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Changes in cognitive function | 24 to 36 months
  Assesment by Montreal Cognitive Assessment questionnaire (MOCA). Minimum value is 0 and maximum value is 30. A higher or equal value to 26 points will be considered normal.

SECONDARY OUTCOMES:
LDL-cholesterol values | 24 to 36 months
  LDL-cholesterol changes will be assessed during the study by routine sample tests (mg/dL)
Changes in Quality of life | 24 to 36 months
  By using the questionnaire called EuroQol EQ-5D-3L assessment. It has 2 parts, the first one has 5 questions with 3 possible answers (5 dimensions and 3 levels), so each health status has a rate called EVA from 1,0000 (the highest value) to - 0,5095 (the worst health status).
  The second part is a visual self-assessment between 0 (the worst health status) and 100 (the best health status). https://euroqol.org/
Direct costs | 24 to 36 months
  Direct costs related with treatments and consultations (€)

OTHER OUTCOMES:
Total Cholesterol | 24 to 36 months
  Total cholesterol evolution during the study in mg/dL
Lp(a) | 24 to 36 months
  Lp(a) evolution during the study in mg/dL
Cost-effectiveness | 24 to 36 months
  €/QUALY

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Hospital de Virxen da Xunqueira de Cee, Cee, A Coruña
  - Hospital Arquiteto Marcide de Ferrol, Ferrol, A Coruña
  - Hospital del Barbanza, Ribeira, A Coruña
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Público da Mariña de Burela, Burela de Cabo, Lugo
  - Hospital de Monforte, Monforte de Lemos, Lugo
  - Hospital do Barco de Valdeorras, O Barco de Valdeorras, Ourense
  - Hospital Alvaro Cunqueiro de Vigo, Vigo, Pontevedra
  - Complejo Hospitalario Universitario de A Coruña, A Coruña
  - Hospital Lucus-Augusti de Lugo, Lugo
  - Complejo Hospitalario Universitario de Ourense, Ourense
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Giugliano RP, Mach F, Zavitz K, Kurtz C, Im K, Kanevsky E, Schneider J, Wang H, Keech A, Pedersen TR, Sabatine MS, Sever PS, Robinson JG, Honarpour N, Wasserman SM, Ott BR; EBBINGHAUS Investigators. Cognitive Function in a Randomized Trial of Evolocumab. N Engl J Med. 2017 Aug 17;377(7):633-643. doi: 10.1056/NEJMoa1701131. PMID 28813214
- [Background] Schwartz GG, Steg PG, Szarek M, Bhatt DL, Bittner VA, Diaz R, Edelberg JM, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Lecorps G, Mahaffey KW, Moryusef A, Pordy R, Quintero K, Roe MT, Sasiela WJ, Tamby JF, Tricoci P, White HD, Zeiher AM; ODYSSEY OUTCOMES Committees and Investigators. Alirocumab and Cardiovascular Outcomes after Acute Coronary Syndrome. N Engl J Med. 2018 Nov 29;379(22):2097-2107. doi: 10.1056/NEJMoa1801174. Epub 2018 Nov 7. PMID 30403574
- [Background] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224
- [Background] Kolodziejczak M, Navarese EP. Role of PCSK9 antibodies in cardiovascular disease: Critical considerations of mortality and neurocognitive findings from the current literature. Atherosclerosis. 2016 Apr;247:189-92. doi: 10.1016/j.atherosclerosis.2016.02.011. Epub 2016 Feb 15. PMID 26926598
- [Background] Lipinski MJ, Benedetto U, Escarcega RO, Biondi-Zoccai G, Lhermusier T, Baker NC, Torguson R, Brewer HB Jr, Waksman R. The impact of proprotein convertase subtilisin-kexin type 9 serine protease inhibitors on lipid levels and outcomes in patients with primary hypercholesterolaemia: a network meta-analysis. Eur Heart J. 2016 Feb 7;37(6):536-45. doi: 10.1093/eurheartj/ehv563. Epub 2015 Nov 17. PMID 26578202
- [Background] Shibata N, Ohnuma T, Higashi S, Higashi M, Usui C, Ohkubo T, Watanabe T, Kawashima R, Kitajima A, Ueki A, Nagao M, Arai H. No genetic association between PCSK9 polymorphisms and Alzheimer's disease and plasma cholesterol level in Japanese patients. Psychiatr Genet. 2005 Dec;15(4):239. doi: 10.1097/00041444-200512000-00004. No abstract available. PMID 16314752
- [Background] Xue-Shan Z, Juan P, Qi W, Zhong R, Li-Hong P, Zhi-Han T, Zhi-Sheng J, Gui-Xue W, Lu-Shan L. Imbalanced cholesterol metabolism in Alzheimer's disease. Clin Chim Acta. 2016 May 1;456:107-114. doi: 10.1016/j.cca.2016.02.024. Epub 2016 Mar 2. PMID 26944571
- [Background] Banach M, Rizzo M, Nikolic D, Howard G, Howard V, Mikhailidis D. Intensive LDL-cholesterol lowering therapy and neurocognitive function. Pharmacol Ther. 2017 Feb;170:181-191. doi: 10.1016/j.pharmthera.2016.11.001. Epub 2016 Nov 16. PMID 27865998
- [Background] Paquette M, Saavedra YGL, Poirier J, Theroux L, Dea D, Baass A, Dufour R. Loss-of-Function PCSK9 Mutations Are Not Associated With Alzheimer Disease. J Geriatr Psychiatry Neurol. 2018 Mar;31(2):90-96. doi: 10.1177/0891988718764330. Epub 2018 Mar 21. PMID 29562810
- [Background] Robinson JG, Rosenson RS, Farnier M, Chaudhari U, Sasiela WJ, Merlet L, Miller K, Kastelein JJ. Safety of Very Low Low-Density Lipoprotein Cholesterol Levels With Alirocumab: Pooled Data From Randomized Trials. J Am Coll Cardiol. 2017 Feb 7;69(5):471-482. doi: 10.1016/j.jacc.2016.11.037. PMID 28153102
- [Background] Seijas-Amigo J, Rodriguez-Penas D, Estany-Gestal A, Suarez-Artime P, Santamaria-Cadavid M, Gonzalez-Juanatey JR. Observational multicentre prospective study to assess changes in cognitive function in patients treated with PCSK9i. Study protocol. Farm Hosp. 2021 Mar 5;45(3):150-154. doi: 10.7399/fh.11569. PMID 33941059
- [Background] Seijas-Amigo J, Gayoso-Rey M, Mauriz-Montero MJ, Suarez-Artime P, Casas-Martinez A, Dominguez-Guerra M, Gonzalez-Freire L, Estany-Gestal A, Codero-Fort A, Rodriguez-Manero M, Gonzalez-Juanatey JR; e investigadores MEMOGAL. Impact of the COVID-19 pandemic in the lipid control of the patients that start PCSK9 inhibitors. Clin Investig Arterioscler. 2022 Sep-Oct;34(5):245-252. doi: 10.1016/j.arteri.2022.01.003. Epub 2022 Feb 3. English, Spanish. PMID 35287972
- [Derived] Seijas-Amigo J, Mauriz-Montero MJ, Suarez-Artime P, Gayoso-Rey M, Reyes-Santias F, Estany-Gestal A, Casas-Martinez A, Gonzalez-Freire L, Rodriguez-Vazquez A, Perez-Rodriguez N, Villaverde-Pineiro L, Castro-Rubinos C, Espino-Paisan E, Cordova-Arevalo O, Rodriguez-Penas D, Cardeso-Paredes B, Ribeiro-Ferreiro M, Rodriguez-Manero M, Cordero A, Gonzalez-Juanatey JR, Memogal Investigators. Cost-Utility Analysis of PCSK9 Inhibitors and Quality of Life: A Two-Year Multicenter Non-Randomized Study. Diseases. 2024 Oct 5;12(10):244. doi: 10.3390/diseases12100244. PMID 39452487
- [Derived] Seijas-Amigo J, Mauriz-Montero MJ, Suarez-Artime P, Gayoso-Rey M, Estany-Gestal A, Casas-Martinez A, Gonzalez-Freire L, Rodriguez-Vazquez A, Perez-Rodriguez N, Villaverde-Pineiro L, Castro-Rubinos C, Espino-Faisan E, Rodriguez-Manero M, Cordero A, Gonzalez-Juanatey JR; Investigadores MEMOGAL. Cognitive Function with PCSK9 Inhibitors: A 24-Month Follow-Up Observational Prospective Study in the Real World-MEMOGAL Study. Am J Cardiovasc Drugs. 2023 Sep;23(5):583-593. doi: 10.1007/s40256-023-00604-6. Epub 2023 Aug 23. PMID 37612529